CLINICAL TRIAL: NCT01718847
Title: Phase II Exploratory Trial to Evaluate the Efficacy and Safety of NOV120101 (Poziotinib) in Lung Adenocarcinoma Patients With Acquired Resistance to 1st Generation EGFR Tyrosine Kinase Inhibitors
Brief Title: NOV120101 Phase 2 Study in NSCLC Patients With Aquired Resistance to 1st Generation EGFR Tyrosine Kinase Inhibitors
Acronym: NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National OncoVenture (Other)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV120101-202
Record Dates: First submitted 2012-10-22; First posted 2012-10-31 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Increased Drug Resistance
Keywords: EGFR Tyrosine Kinase Inhibitor; Aquired resistance to EGFR TKI; Pan-Her inhibitor
MeSH Terms: interventions — HM781-36B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NOV120101 (Poziotinib) (Experimental): 16 mg PO once daily until disease progression or unacceptable toxicity development
  Interventions: Drug: NOV120101 (Poziotinib)

INTERVENTIONS:
Drug: NOV120101 (Poziotinib) — 16 mg PO once daily until disease progression or unacceptable toxicity development
  Other Names: HM781-36B

SUMMARY:
The purpose of this open-label, single-arm, multi-center phase II trial is to evaluate the efficacy and safety of novel pan-HER inhibitor, NOV120101 (Poziotinib), as a 2nd line monotherapy agent in lung adenocarcinoma patients with acquired resistance to prior EGFR tyrosine kinase inhibitors (TKIs).

DETAILED DESCRIPTION:
Acquired resistance to prior EGFR TKIs is considered as "unmet medical need" in clinical practice. To evaluate the efficacy of NOV120101 (Poziotinib) as a second-line monotherapeutic agent, patients with acquired resistance to gefitinib or erlotinib will be enrolled in this study. Subjects will receive NOV120101 (Poziotinib) 16 mg PO once daily until disease progression or unacceptable toxicity development. Progression free survival (PFS) will be analyzed as the primary endpoint in this trial. Secondary endpoints including PFS rate at 16 weeks, ORR and DCR will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 20 years or older
2. Pathologically confirmed stage IIIB (unresectable) or IV lung adenocarinoma
3. Patients who have 1 or more than 1 measurable or evaluable but unmeasurable lesions according to RECIST ver1.1
4. Patients who received prior 1st generation EGFR TKIs (gefitinib or erlotinib) monotherapy and meet the following criteria:

   1. Patients with EGFR mutation (e.g., G719X, exon 19 deletion, L858R, L861Q, etc) known to be associated with sensitivity to TKIs
   2. Patients who showed objective clinical benefit from treatment with an EGFR TKI as defined by either:

      * Patients who showed complete (CR) or partial response (PR), or
      * Patients who maintained stable disease (SD) status ≥ 6 months
   3. Patients who showed progressive disease (PD, RECIST ver1.1) while on continuous treatment with gefitinib or erlotinib within the last 30 days (However, patients whose progressive disease is limited in the brain cannot participate in this trial.)
   4. No intervening systemic chemotherapy between cessation of the EGFR TKI and participation of this study
5. Patients who agree to the collection of tumor tissue specimen
6. ECOG performance status ≤ 2
7. Life expectancy of ≥ 12 weeks
8. Adequate hematological, hepatic and renal functions:

   WBC ≥ 4,000/mm3, Platelet ≥ 100,000/mm3, Serum creatinine ≤ 1.5 X ULN, AST and ALT ≤ 2.5 X ULN, Total bilirubin ≤ 1.5 X ULN
9. Patients who give written informed consent voluntarily

Exclusion Criteria:

1. Patients who receive IP within 3 days from prior treatment with gefitinib or erlotinib
2. NCI-CTCAE grade > 1 adverse events due to treatment with gefitinib or erlotinib
3. Prior systemic chemo, immuno, hormonal and/or biological therapy except gefitinib or erlotinib within 4 weeks before IP administration
4. Acquired resistance to EGFR TKI due to conversion of adenocarcinoma into small cell lung cancer
5. Patients who received major surgery within 4 weeks before IP administration
6. Symptomatic CNS metastases (patients with radiologically and neurologically stable metastases and being off corticosteroids for at least 4 weeks are able to participate in this trial.)
7. History of other malignancies except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for ≥ 3 years and considered to be cured by investigator's judgment
8. Known pre-existing interstitial lung disease (ILD)
9. NYHA class III or IV heart failure, uncontrolled hypertension, unstable angina or myocardial infarction within 6 months, poorly controlled arrhythmia or other clinically significant cardiovascular abnormalities at investigator's discretion
10. Patients whose left ventricle ejection fraction (LVEF) is below the institutional lower limit of normal (if no lower limit of normal is defined in the site, the lower limit is 50%.)
11. Patients with known active hepatitis B, HIV infection, or other uncontrolled infectious disease
12. Clinically significant or recent acute gastrointestinal disorders with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption disorders, CTCAE grade ≥ 2 diarrhea due to any etiology)
13. Patients who cannot receive IP by mouth and be diagnosed with clinically significant gastrointestinal disorders which can prevent administration, transit or absorption of the IP
14. Pregnancy or breast-feeding
15. Women of childbearing potential (WOCBP) or men who are unwilling to use adequate contraception or be abstinent during the trial and for at least 2 months after the end of treatment
16. Patients who received other investigational products except gefitinib and erlotinib within 4 weeks before participation
17. Patients who cannot participate in this trial by investigator's judgment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | By 1 year after enrollment of the last subject
  The length of time during and after medication or treatment during which the disease being treated (usually cancer) does not get worse.

SECONDARY OUTCOMES:
PFS rate at 16 weeks | 16 weeks
  The proportion of Patients maintaining progress-free status at 16 weeks
Objective response rate (ORR) | By 1 year after enrollment of the last subject
  The proportion of patients with partial response or complete response at their best tumor treatment evaluation
Disease control rate (DCR) | By 1 year after enrollment of the last subject
  The proportion of patients with CR, PR and/or stable disease (SD)
Overall survival (OS) | By 1 year after enrollment of the last subject
Time to progression (TTP) | By 1 year after enrollment of the last subject
Time to objective response | By 1 year after enrollment of the last subject
Duration of objective response | By 1 year after enrollment of the last subject
Duration of disease control | By 1 year after enrollment of the last subject
Change of quality of life (QoL) measured by EQ-5D questionnaire | baseline and the end of treatment, by 1 year after enrollment of the last subject

OTHER OUTCOMES:
Population pharmacokinetics (PK) of NOV120101 (Poziotinib) | By 3 months after enrollment of the last subject
  The study of the sources and correlates of variability in drug concentrations among individuals who are the target patient population receiving clinically relevant doses of a study drug. Certain patient demographic, pathophysiological, and therapeutical features, such as body weight, excretory and metabolic functions, and the presence of other therapies, can regularly alter dose-concentration relationships.
Subgroup analyses with the genetic information | by 1 year after enrollment of the last patient
  Subgroup analysis, in the context of design and analysis of study drug, refers to looking for pattern in a subset of the subjects according to genotype

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Youn Han, MD. Ph.D, Study Chair — National Cancer Center, Goyang-si, Gyeonggi-do, Republic of Korea,Asan Medical Center, Songpa-gu, Seoul, Republic of Korea,; Ki Hyeong Lee, MD, Ph.D, Principal Investigator — Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk-do, Republic of Korea; Sang-We Kim, MD, Ph.D, Principal Investigator — Asan Medical Center, Songpa-gu, Seoul, Republic of Korea; Young Joo Min, MD, Ph.D, Principal Investigator — Ulsan University Hospital, Dong-gu, Ulsan, Republic of Korea; Eunkyung Cho, MD, Ph.D, Principal Investigator — Gachon University Gil Medical Center, Incheon, Republic of Korea
Locations (5):
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Asan Medical Center, Songpa-gu, Seoul
  - Ulsan University Hospital, Dong-gu, Ulsan
  - Gachon University Gil Medical Center, Incheon